CLINICAL TRIAL: NCT01333306
Title: Enhancing Cognitive Training Using tDCS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: University of New South Wales, University of New South Wales
Purpose: Basic Science
Other Study IDs: 10269
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2010-09

CONDITIONS: Cognition
Keywords: tDCS; cognitive training
MeSH Terms: interventions — Transcranial Direct Current Stimulation

ARMS (1):
- tDCS and cognitive training (Experimental)
  Interventions: Procedure: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Procedure: Transcranial direct current stimulation (tDCS)

SUMMARY:
Cognitive rehabilitation involves enhancing an individual's capacity to process information to improve their everyday functioning. One common form of intervention is computerised cognitive training (CT); however, efficacy results have been mixed. This research aims to investigate a novel method for enhancing outcomes from CT through combining CT with transcranial direct current stimulation (tDCS), a non-invasive and painless form of brain stimulation. In this study we aim to determine the efficacy of this approach through comparing in a randomized controlled study tDCS combined with CT versus CT and tDCS alone in healthy participants. We hypothesise that tDCS combined with CT will have greater generalisability effects than the other conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy right-handed subjects aged 18 to 40

Exclusion Criteria:

* Concurrent medication likely to affect mental performance
* History of drug or alcohol abuse or dependence current or in the last 3 months
* Any psychiatric or neurological disorder, recent head injury, or history of seizure or stroke

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2010-09; Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute Building, Sydney, New South Wales, Australia